CLINICAL TRIAL: NCT02206347
Title: The Effect of Prioritization of Attentional Allocation on Postural-suprapostural Tasking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201209056RIC
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Attention on Posture; Attention on Supraposture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- attention focus (Other)
  Interventions: Behavioral: attention focus

INTERVENTIONS:
Behavioral: attention focus

SUMMARY:
Postural-suprapostural task is defined as postural control takes place while at least one other concurrent task is being performed, and appropriate locus of attentional allocation is considered a critical factor for successful postural-suprapostural execution. Recent studies have indicated that the behavior performance of postural-suprapostural task would be affected by the prioritization of attentional allocation (postural-first vs. suprapostural-first); however, the inference of the appropriateness of attention prioritization is primarily limited to behavior observations and lacks direct neural evidences. How the effect of attentional priority between postural and suprapostural tasks on postural-suprapostural performance and its underlying cortical mechanism is rarely understood. By adopting postural-first and suprapostural-first strategies for postural-suprapostural task, the purpose of this 2-year research project is to 1) investigate the differences in performance quality and intrinsic neural mechanisms effect of a postural-suprapostural task for healthy adults with the analysis of event-related potential (ERP) and non-linear dynamics of behavior measures; 2) investigate brain plastic changes and the appropriateness of strategy use. In the first year, the attention prioritization effect on reciprocity of a postural-suprapostural task will be characterized by integrating the results of behavior performance and ERP causal connectivity with a special focus on validation of prevailing theoretical models. In the second year, the difference of task fluent for learning a postural-suprapostural task with postural-first/suprapostural-first strategy will be studied through the spatial and time variations in alpha rhythm after principle component analysis. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of concurrent postural and motor suprapostural tasks, but to optimize treatment strategy for patients with balance or multi-tasking disturbances.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults without neuromuscular / cardiovascular disease

Exclusion Criteria:

* pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
precision-grip force error | up to 2 years
  The precision-grip force error is used as the performance of suprapostural task
balance | up to 2 years
  The balance measure is used as the postural performance.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan